CLINICAL TRIAL: NCT03143959
Title: A Prospective Study of the Impact of Abdominoplasty on the Symptoms of Back Pain and Urinary Incontinence in the Post Partum Population.
Brief Title: Functional Improvement With Abdominoplasty
Status: Completed | Type: Observational
Sponsor: The Caps Clinic (Other)
Responsible Party: Principal Investigator, Alastair Taylor, Plastic Surgeon, The Caps Clinic
Other Study IDs: FuncAbdo
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Lower Back Pain Chronic; Urinary Incontinence; Recti Diastasis; Abdominoplasty
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study investigates the impact of abdominoplasty in the post partum population on the symptoms of back pain and urinary incontinence. Patients presenting for abdominoplasty fill out validated questionnaires for both back pain (Oswestry Disability Index) and urinary incontinence (ICIQ-UI short form). They complete the same questionnaires 6 weeks and 6 months post op. The prospectively gathered data gives an insight into the incidence of functional symptoms in this post partum group preop as well as the degree of improvement gained postop. This is a multicenter trial with 9 surgeons submitting patients to the study, which ran for 19 months.

DETAILED DESCRIPTION:
Abdominoplasty has long been considered a cosmetic procedure, improving the shape of the abdomen by excess skin removal, liposuction and rectus muscle plication. Performed chiefly on the post-partum and weight loss population, there have been reports of improvement in the functional symptoms of back pain and incontinence following abdominoplasty with rectus plication but there has been no prospective multicentre study to investigate the issue.

The incidence of chronic back pain greater than two years following pregnancy has been reported between 5% to 21.1%. Persistent urinary incontinence rates 10 to 12 years after pregnancy range between 25% to 37.9%. Vaginal delivery is associated with a higher incidence of long term stress incontinence. The Australian female population is approximately 11m. With a 24% rate of childlessness up to 1.67m Australian women are suffering chronic back pain and 3.2m stress incontinence. Both these conditions negatively affect the quality of life and are usually under reported.

This is a multicentre prospective study on the impact of abdominoplasty on back pain and urinary incontinence in the post-partum population. All post-partum patients presenting for abdominoplasty were enrolled to give an indication of incidence of symptoms in this population as well as the magnitude of improvement or deterioration.

The prospective study utilised validated questionnaires. For back pain the Oswestry Disability Index (ODI) was selected as it is an excellent measure of a patient's functional disability and has been in use for nearly 40 years. The Index is a multiple choice questionnaire, divided into 10 sections assessing Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Social Life, Travelling and the impact on Employment and House making. Each section is scored from 0 to 5, the maximum score is 50. The score is then doubled to become a percentage disability index. Urinary Incontinence was measured with the International Consultation On Incontinence Questionnaire - Urinary Incontinence - Short Form (ICIQ-UI-SF). This is also a multiple-choice questionnaire asking the patient to score the frequency of urine leakage, how much they think leaks and on a scale of one to ten how much it interferes with daily life. It is not a disability index like the Oswestry. A maximum score is 21 with urine leaking all the time, large amounts and interfering with life a great deal.

Patients completed the questionnaires pre abdominoplasty and at 6 weeks and 6 months post operation. Demographic information was collected; Age, Parity, Age Range of Children (the years between the oldest and youngest), Method of Birth (Vaginal or Caesarean) and BMI preoperatively. Surgical data was also obtained; Method of Abdominoplasty, Weight Removed, Volume of Liposuction, Width of Diastasis and the presence of a Hernia. No data on postoperative complications was collected. Patients signed an informed consent form to participate after reading an information pamphlet and the study was approved by the ACT Health Human Research Ethics Committee.

A presentation at the 37th Annual Australasian Society of Aesthetic Plastic Surgeons conference in August 2014 recruited surgeons to the study. Nine surgeons agreed to take part and were given packs of questionnaires, patient information brochures, consent forms, demographic forms and a surgeons information sheet. The nine participants were individual private practitioners, four from Sydney NSW and one each from Canberra ACT, Toowoomba QLD, Brisbane QLD, Gold Coast QLD and Newcastle NSW, a mix of capital city and smaller regional centres along the east coast of Australia.

The objective was to study both the incidence of functional symptoms in the population presenting for abdominoplasty as well as the outcome. Study surgeons were instructed to enrol all post-partum abdominoplasty patients. Nulliparous weight loss patients were excluded as were males. The completed forms were posted back to the study author who compiled the results. Statistical analysis was performed by Datalytics (Bruce ACT).

ELIGIBILITY:
Inclusion Criteria:

* Post Partum Females presenting for abdominoplasty

Exclusion Criteria:

* Males and non post partum females presenting for abdominoplasty

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any post partum female presenting for abominoplasty regardless of whether they have functional symptoms or not.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Back pain | 6 months
  Reduction in back pain following abdominoplasty measured by questionnaire
Urinary incontinence | 6 months
  reduction in urinary incontinence following abdominoplasty measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Taylor, FRACS, Principal Investigator — The Caps Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noren L, Ostgaard S, Johansson G, Ostgaard HC. Lumbar back and posterior pelvic pain during pregnancy: a 3-year follow-up. Eur Spine J. 2002 Jun;11(3):267-71. doi: 10.1007/s00586-001-0357-7. Epub 2001 Dec 8. PMID 12107796
- [Background] Ostgaard HC, Zetherstrom G, Roos-Hansson E. Back pain in relation to pregnancy: a 6-year follow-up. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2945-50. doi: 10.1097/00007632-199712150-00018. PMID 9431631
- [Background] To WW, Wong MW. Factors associated with back pain symptoms in pregnancy and the persistence of pain 2 years after pregnancy. Acta Obstet Gynecol Scand. 2003 Dec;82(12):1086-91. doi: 10.1046/j.1600-0412.2003.00235.x. PMID 14616251
- [Background] Altman D, Ekstrom A, Gustafsson C, Lopez A, Falconer C, Zetterstrom J. Risk of urinary incontinence after childbirth: a 10-year prospective cohort study. Obstet Gynecol. 2006 Oct;108(4):873-8. doi: 10.1097/01.AOG.0000233172.96153.ad. PMID 17012448
- [Background] Viktrup L, Rortveit G, Lose G. Risk of stress urinary incontinence twelve years after the first pregnancy and delivery. Obstet Gynecol. 2006 Aug;108(2):248-54. doi: 10.1097/01.AOG.0000226860.01127.0e. PMID 16880292
- [Background] MacArthur C, Wilson D, Herbison P, Lancashire RJ, Hagen S, Toozs-Hobson P, Dean N, Glazener C; Prolong study group. Urinary incontinence persisting after childbirth: extent, delivery history, and effects in a 12-year longitudinal cohort study. BJOG. 2016 May;123(6):1022-9. doi: 10.1111/1471-0528.13395. Epub 2015 Apr 2. PMID 25846816
- [Background] 7. Australian Bureau of Statistics 2000, Births, Australia, 2000, cat no. 3301.0, ABS, Canberra
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Davidson M, Keating JL. A comparison of five low back disability questionnaires: reliability and responsiveness. Phys Ther. 2002 Jan;82(1):8-24. doi: 10.1093/ptj/82.1.8. PMID 11784274
- [Background] Timmermans L, Falez F, Melot C, Wespes E. Validation of use of the International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF) for impairment rating: a transversal retrospective study of 120 patients. Neurourol Urodyn. 2013 Sep;32(7):974-9. doi: 10.1002/nau.22363. Epub 2012 Dec 31. PMID 23281067